CLINICAL TRIAL: NCT03588039
Title: Phase 1 Study With Expansion Cohorts to Assess the Safety, Tolerability, and Activity of Oraxol (Paclitaxel + HM30181A) in Combination With Pembrolizumab in Subjects With Advanced Solid Malignancies
Brief Title: Study of Oraxol and Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to lack of funding
Sponsor: Athenex, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-011; KEYNOTE-E06 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2018-06-13; First posted 2018-07-17 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose escalation-Arm 1 (Experimental): During the dose escalation period Oraxol will be administered once daily for 2 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose escalation-Arm 2 (Experimental): During the dose escalation period Oraxol will be administered once daily for 3 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose escalation-Arm 3 (Experimental): During the dose escalation period Oraxol will be administered once daily for 4 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose escalation-Arm 4 (Experimental): During the dose escalation period Oraxol will be administered once daily for 5 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose escalation-Arm 5 (Experimental): During the dose escalation period Oraxol will be administered once daily for 5 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose escalation-Arm 6 (Experimental): During the dose escalation period Oraxol will be administered once daily for 5 days per week for 2 weeks followed by 1 week off treatment (2 weeks on and 1 week off). Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose expansion-Gastric/GE (Experimental): The dose expansion period will enroll subjects with gastric/gastro-esophageal cancer to further evaluate the activity and safety of the study treatment. Oraxol will be administered at the dose determined from part 1 for 2 out of 3 weeks. Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab
- Dose expansion-NSCLC cancer (Experimental): The dose expansion period will enroll subjects with NSCLC to further evaluate the activity and safety of the study treatment. Oraxol will be administered at the dose determined from part 1 for 2 out of 3 weeks. Pembrolizumab will be administered on Day 1 of each 3-week cycle.
  Interventions: Drug: Oraxol; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Oraxol — Oral paclitaxel will be supplied in capsules and oral HM30181AK-US will be supplied in tablets
  Other Names: oral HM30181A + oral paclitaxel
Biological: Pembrolizumab — Intravenously administered
  Other Names: Keytruda

SUMMARY:
This is an open-label, Phase 1 dose-escalation study followed by a 2-arm expansion cohort of Oraxol administered in combination with pembrolizumab.

DETAILED DESCRIPTION:
This is a two part study. The dose escalation part will enroll subjects with advanced solid tumors for which pembrolizumab is an FDA-approved therapy, to determine the MTD and identify the recommended phase 2 dose of paclitaxel administered as Oraxol in combination with pembrolizumab. Upon determination of the phase 2 dose, the dose expansion part will enroll subjects with advanced/metastatic gastric/gastro-esophageal, or NSCLC into 2 independent cohorts/arms to further evaluate the activity and safety of the study treatment.

ELIGIBILITY:
Inclusion Criteria

Eligible subjects must have/be:

* Able to understand and sign an informed consent form
* Age ≥18 years
* Dose Escalation: Histologically confirmed metastatic or unresectable solid tumors for which pembrolizumab is an FDAapproved therapy
* Dose Expansion: Histologically confirmed diagnosis of advanced or metastatic NSCLC or gastric/gastro-esophageal adenocarcinoma:

NSCLC:

* Subjects with actionable mutations or alterations must have progressed on prior FDA approved therapy for these aberrations.
* Subjects must have progressed on a prior FDA-approved single agent immunotherapy (antiPD1/anti-PD-L1) in first line (1L) or progressed on a prior FDA approved immunotherapy + chemotherapy combination therapy in 1L, as long as the chemotherapy did not include a taxane.

Gastric/Gastro-esophageal

* Histologically confirmed diagnosis of advanced or metastatic gastric/gastro-esophageal adenocarcinoma or esophageal squamous cell carcinoma.
* Subjects must have progressed on previous anti-PD-1 therapy as single agent or combination therapy.
* Must have at least one measurable site of disease as defined as per RECIST v1.1 criteria
* ECOG Performance Status ≤1
* The following laboratory values obtained ≤14 days prior to Cycle 1/Day 1 dosing:
* Absolute neutrophil count (ANC) ≥1.5 x 109/L
* Platelet count ³100 x 109/L
* Hemoglobin ≥9.0 g/dL
* Total and direct bilirubin within normal range
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) £3 x upper limit of normal (ULN)
* Gamma-glutamyl transferase (GGT) ≤5 x ULN
* Alkaline phosphatase ≤3 x ULN or ≤5 x ULN if bone or liver metastasis is present
* Serum creatinine £2 x ULN, or 24-hr urine creatinine clearance calculation ³ 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) ≤1.5 x ULN OR if a subject is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants for 7 days prior to receiving study treatment
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* No concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder
* Subjects receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
* Men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) OR agree to use a condom with spermicide and to not donate sperm during the study and for at least 30 days following last dose of Oraxol
* Female subjects must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of assigned study treatment. Abstinence is also an acceptable form of contraception.
* Subjects who are of childbearing potential must have a negative serum pregnancy test at Screening and within 96 hours before Week 1 dosing.
* Willing to return for follow-up
* Willing to provide blood samples for correlative research purposes
* Life expectancy of at least 3 months

Exclusion Criteria

* Eligible subjects must not have/be:
* Subjects with history of prior treatment with taxanes (eg, paclitaxel, docetaxel, cabazitaxel) in expansion cohorts only
* History of prior significant toxicity from anti-PD-1 or anti-PD-L1 therapy requiring discontinuation of treatment
* Subjects who have received recent anti-cancer therapy defined by:
* Chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosurea, mitomycin-C, targeted therapy, and radiation) ≤28 days prior to starting study drug, or who have not recovered from side effects of such therapy
* Last administration of nitrosurea or mitomycin-C ≤42 days prior to starting study drug, or who have not recovered from the side effects of such therapy
* Targeted therapy (eg, sunitinib, sorafenib, pazopanib) ≤14 days prior to starting study drug, or who have not recovered from the side effects of such therapy; or
* Radiotherapy ≤28 days prior to starting study drug, or ≤14 days prior to starting study drug in the case of localized radiotherapy (eg, for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of pembrolizumab. The following are exceptions to this criterion: Intranasal, inhaled, topical corticosteroids, or local corticosteroid, injections (eg, intra-articular injection), systemic corticosteroids at doses not to exceed 10 mg/day of prednisone or its equivalent.
* Vaccinated with live, attenuated vaccines within 28 days of the first dose of the study drug
* Active or prior documented autoimmune or inflammatory disorders (including but not limited to inflammatory bowel disease [eg, colitis, Crohn's disease], celiac disease, or other serious gastrointestinal (GI) chronic conditions associated with diarrhea; type 1 diabetes mellitus; multiple sclerosis; systemic lupus erythematosus; Wegener's granulomatosis; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis; uveitis; etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:
* Subjects with vitiligo or alopecia
* Subjects with hypothyroidism (eg, following Hashimoto's thyroiditis) stable on hormone replacement therapy or psoriasis not requiring systemic treatment
* Subject has impairment of GI function or GI disease that may significantly alter the absorption of study drugs (including gastric bypass surgery and total gastrectomy). Subjects with partial gastrectomy may be included in the trial.
* Subjects who have undergone major surgery (eg, intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤28 days prior to starting study treatment, or subjects who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤7 days prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Uncontrolled concurrent illness, including but not limited to ongoing or active serious infection requiring systemic antimicrobials (within 14 days prior to first dose of Oraxol), arterial hypertension (>160/100 mm/Hg on antihypertensive medications), uncontrolled endocrine diseases, altered mental status or psychiatric illness/social situations that would limit compliance with protocol requirements and/or obscure study results.
* Known or suspected diagnosis of human immunodeficiency virus (HIV) or chronic active Hepatitis B or C, or cirrhosis.
* Clinically significant pulmonary illness resulting in Grade ≥2 hypoxia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE, v4.03]) or any requirement for supplemental oxygen, or pulse oximetry less than 90% saturation on room air
* Symptomatic or uncontrolled brain metastases requiring current treatment (less than 28 days from last cranial radiation or 28 days from last steroids use).
* Impaired cardiac function or clinically significant cardiac disease including the following:
* Clinically significant arrhythmias (except chronic well controlled atrial fibrillation)
* New York Heart Association (NYHA) Class III or IV congestive heart failure
* Angina pectoris ≤6 months
* Myocardial infarction within the last 12 months
* Subjects with a healing or open wound
* Lack of recovery of prior AEs to Grade ≤1 severity (NCI CTCAE v4.03) (except alopecia) due to medications administered prior to the first dose of the trial drugs.
* Any other condition or finding (including social situation) that in the opinion of the Investigator may render the patient at excessive risk for treatment complications or may not be able provide evaluable outcome information.
* Pregnant or breast-feeding women
* Known allergy to any of the formulation components of Oraxol (oral paclitaxel or HM30181A) or pembrolizumab
* Currently taking following prohibited concomitant medication:
* Medication known to be strong inhibitors (gemfibrozil) or inducers (rifampin) of cytochrome P450 (CYP)2C8. Subjects who are currently taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication 14 days before dosing and remain off that medication during treatment with Oraxol.
* Strong CYP3A4 inducer (eg, rifampin or St. John's Wort) or a strong CYP3A4 inhibitors (eg, ketoconazole) or a moderate CYP3A4 inhibitor including neurokinin 1 (NK1) inhibitors (eg, aprepitant and rolapitant) within 14 days prior to treatment administration
* Medication known to be strong P-gp inhibitors or inducers. Subjects who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication 7 days before dosing and remain off that medication during treatment with Oraxol.
* An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg, digoxin, dabigatran) within 1 day prior to start of Oraxol dosing in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Determination of MTD | 3 weeks
  dose limiting toxicities occuring in the first cycle of therapy
Tumor response rate | 24 months
  Proportion of subjects in each arm and part 2 with confirmed tumor response

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
  To determine the progression free survival after initiation of treatment with Oraxol in subjects
Overall survival (OS) | 24 months
  To determine the overall survival after initiation of treatment with Oraxol in subjects
Duration of response (DOR) | 24 months
  The duration of response will be measured in subjects associated with Oraxol administered in combination with pembrolizumab in subjects with advanced/metastatic gastric/gastro-esophageal, or NSCLC who have stable disease or progressed on previous anti-PD1 or anti-PDL1 therapy
Pharmacokinetics of Oraxol | Day 1 and day 2
  Plasma concentrations of Oraxol
Disease Control Rate (DCR) | 24 months
  The disease control rate, defined as the proportion of subjects whose best response is complete response (CR), partial response (PR), or stable disease (SD) divided by the total number of evaluable subjects in each cohort.
Incidence of Adverse Events | 24 months
  The incidence of Treatment Emergent Adverse Events and Treatment-related Adverse Events will be summarised using descriptive statistics.
Time to response | 24 months
  To determine the time to response, defined as the time from the treatment initiation to first documented response

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Sr. Vice President of Clinical Development
Locations (4):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No